CLINICAL TRIAL: NCT04184960
Title: Performance of Endoscopic and Histological Criteria of Atrophic Gastritis and Intestinal Metaplasia in Predicting Risk of Gastric Cancer - a Multicenter Case Control Study
Brief Title: AG & IM in CA Stomach Protocol
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Hon Chi Yip, Associate Consultant, Chinese University of Hong Kong
Other Study IDs: CRE-2019.341
Record Dates: First submitted 2019-12-01; First posted 2019-12-04 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Gastric Cancer; Atrophic Gastritis; Intestinal Metaplasia
Keywords: Gastric cancer; Gastroscopy; Atrophic gastritis; Intestinal metaplasia
MeSH Terms: conditions — Stomach Neoplasms; Gastritis, Atrophic | interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 4 random biopsies would be taken in specific location of the stomach during gastroscopy. (Lesser curvature mid antrum, greater curvature mid antrum, lesser curvature mid corpus, greater curvature mid corpus)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastric cancer cohort: Cohort of patients with gastric cancer
  Interventions: Diagnostic Test: Gastroscopy and gastric biopsies
- Non-gastric cancer cohort: Cohort of patients without gastric cancer
  Interventions: Diagnostic Test: Gastroscopy and gastric biopsies

INTERVENTIONS:
Diagnostic Test: Gastroscopy and gastric biopsies — Gastroscopy would be performed to assess the degree of atrophic gastritis and intestinal metaplasia. In addition, four random biopsies would be taken in the stomach for histological assessment of AG and IM

SUMMARY:
This is a multi-center prospective case control study aiming to compare different methods of risk stratification models in predicting the risk of gastric cancer development.

DETAILED DESCRIPTION:
The case control study would compare which type of assessment (Endoscopic / histological) is more accurate in predicting the risk of gastric cancer development.

The risk factor assessment would be based on the following criteria.

Endoscopic assessment:

1. Atrophic gastritis, based on Kimura Takemoto Classification
2. Kyoto classification of gastritis
3. Intestinal metaplasia, based on Endoscopic Mapping and Grading of Intestinal Metaplasia (EGGIM) Histological assessment (Based on random biopsies)

1. Operative Links on Gastritis Assessment 2. Operative Links on Gastric Intestinal Metaplasia

ELIGIBILITY:
Two groups of patients would be recruited in this case control study.

1. Gastric neoplasia group Patients with newly diagnosed or history of cancer of stomach or gastric high grade dysplasia.
2. Control group Patients with no prior history of gastric dysplasia or cancer

Inclusion criteria:

1. Age 40 or above
2. Undergo elective upper gastrointestinal endoscopy

Exclusion criteria:

1. Patients with history of gastrectomy
2. Patients with severe thrombocytopenia (Platelet count <50) or coagulopathy (INR > 1.5 or on anticoagulation)
3. Contraindication to upper gastrointestinal endoscopy
4. Allergy towards sedative agents (Midazolam / Diazepam) or local anaesthetic spray (Lignocaine)
5. Patients who cannot give informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with or without gastric cancer undergoing elective endoscopy would be recruited if they fulfil inclusion and exclusion criteria. Subsequently they would be analysed based on "Gastric cancer" and "Non-gastric cancer" cohorts.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-12-05 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Endoscopic grading of atrophic gastritis (Kimura Takemoto Classification) | Cross sectional study, day 0
  Endoscopic description of severity of gastric atrophy
Endoscopic grading of intestinal metaplasia (EGGIM) | Cross sectional study, day 0
  Endoscopic mapping of degree of intestinal metaplasia
Kyoto classification of gastritis | Cross sectional study, day 0
  Descriptive findings of gastritis
Operative links on gastritis assessment (OLGA) | Cross sectional study, day 0
  Biopsy based risk stratification panel based on severity of atrophic gastritis
Operative links on gastric intestinal metaplasia (OLGIM) | Cross sectional study, day 0
  Biopsy based risk stratification panel based on severity of intestinal metaplasia

CONTACTS AND LOCATIONS:
Overall Officials: Hon Chi Yip, Principal Investigator — Chinese University of Hong Kong
Locations (4):
- Prince of Wales Hospital, Hong Kong, Hong Kong
- Osaka International Cancer Institute, Osaka, Japan
- Changi General Hospital, Singapore, Singapore
- King Chulalongkorn Memorial Hospital and Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No